CLINICAL TRIAL: NCT02376075
Title: Effects of Linagliptin on Endothelial- , Renal-, and Retinal Function in Comparison to Placebo in Patients With Hypertension and Albuminuria
Brief Title: Effects of Linagliptin on Endothelial- , Renal-, and Retinal Function in Patients With Hypertension and Albuminuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: Ikfe GmbH (Industry); MLM Medical Labs GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ikfe-Lina-003; 2012-004300-35 (EudraCT Number)
Record Dates: First submitted 2015-02-11; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Arterial Hypertension; Albuminuria
MeSH Terms: conditions — Hypertension; Albuminuria | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, tablets, administered once daily as add on to pre-existing antihypertensive treatment
  Interventions: Drug: Placebo
- Linagliptin (Active Comparator): Linagliptin, tablets containing 5 mg, administered once daily as add on to pre-existing antihypertensive treatment
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — Intake of tablets containing 5 mg Linagliptin, administered once daily as add on to pre-existing antihypertensive treatment for 6 weeks
  Other Names: Trajenta
  Arms: Linagliptin
Drug: Placebo — Intake of Placebo, administered once daily as add on to pre-existing antihypertensive treatment for 6 weeks
  Arms: Placebo

SUMMARY:
A recent study with the DPP-IV inhibitor Linagliptin showed an improvement in the urinary albumin creatinine ratio in patients with diabetic nephropathy. Gutzwiller et. Al. have shown that GLP-1 increases renal Na secretion and inhibits renal H secretion, further indicating some direct renal effects of GLP-1.

Therefore, it seems likely that treatment with the DPP-IV inhibitor Linagliptin evolves several beneficial effects on microvascular and endothelial function beyond glucose control which most probably have an impact on the progression of renal and retinal microvascular disease.

The objective of this trial is to investigate the effect of Linagliptin in comparison to placebo on the UACR in patients with high blood pressure and an increased albumin excretion. Numerous, equivalent endothelial, renal, and retinal parameters serve as objectives of the study. All study parameters will be handled in an exploratory sense for the generation of models to further discuss the role of DPP-IV inhibition on renal and retinal physiology.

DETAILED DESCRIPTION:
Renal tissue damage and an increase in the albumin excretion rate is a strong predictor for the development and progression of endothelial dysfunction and the development of microvascular and/or macrovascular complications. Increased blood pressure as well as increased glucose levels were found to impair renal- and retinal function, and a close association in the incidence and progression rate of retinopathy and nephropathy could be observed. Endothelial dysfunction and alterations in microvascular blood flow are early pathogenetic features in the development of renal and retinal tissue damage as found in patients with arterial hypertension and / or diabetes mellitus. A couple of studies have shown that urinary albumin excretion is associated with morphological and functional alterations in retinal microvascular blood flow. In patients with arterial hypertension blood pressure lowering treatment were shown to decrease the albumin excretion rate and to improve endothelial function of the retinal vasculature.

Recently DPP-IV Inhibitors have been introduced in the treatment of type 2 diabetes mellitus. Beside the metabolic effects of this drug class, several pleiotropic effects beyond metabolic control were documented in numerous studies, and are the topic of ongoing clinical research. Treatment with DPP-IV inhibitors was found to improve myocardial and endothelial function, to improve blood lipids, to lower blood pressure and to improve markers of renal function. GLP-1 receptors in vessels, kidney and the heart might account for those glucose independent effects of GLP-1. However, it is also conceivable that DPP-IV inhibition might exert vascular effects independent from GLP-1. In vitro studies demonstrated that DPP-IV is expressed in endothelial cells, and the inhibition of DPP-IV reduced the microvascular tone through direct mediation of the nitric oxide system. Therefore, it seems conceivable that the glucose independent effects of DPP-IV inhibition might be mediated through GLP-1 receptor signaling and /or direct inhibition of the enzyme DPP-IV in vascular, renal, or retinal cells.

A recent study with the DPP-IV inhibitor Linagliptin showed an improvement in the urinary albumin creatinine ratio in patients with diabetic nephropathy. Gutzwiller et. Al. have shown that GLP-1 increases renal Na secretion and inhibits renal H secretion, further indicating some direct renal effects of GLP-1.

Therefore, it seems likely that treatment with the DPP-IV inhibitor Linagliptin evolves several beneficial effects on microvascular and endothelial function beyond glucose control which most probably have an impact on the progression of renal and retinal microvascular disease.

The objective of this trial is to investigate the effect of Linagliptin in comparison to placebo on the UACR in patients with high blood pressure and an increased albumin excretion. Numerous, equivalent endothelial, renal, and retinal parameters serve as objectives of the study. All study parameters will be handled in an exploratory sense for the generation of models to further discuss the role of DPP-IV inhibition on renal and retinal physiology.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated written informed consent to participate in the trial
* Arterial hypertension
* Stable antihypertensive treatment within the last 3 months
* Age ≥ 45 - ≤ 80 years
* Micro- or macroalbuminuria defined as UACR in morning urine > 20 mg/g in female and > 30 mg/g in male and/or arterial hypertension for more than 5 years currently treated with two or more antihypertensive drugs to control blood pressure and a history of cardiovascular disease or stroke.
* Patient consents that his/her family physician will be informed of trial participation

Exclusion Criteria:

* History of type 1 diabetes
* History of type 2 diabetes
* Uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg)
* Acute infections
* Any history of glomerulonephritis
* Any kidney disease not caused by hypertension as judged by the Investigator
* Glomerular filtration rate (GFR) < 30 ml/min (estimated by use of the Modification of Diet in Renal Disease (MDRD) formula)
* Medical history of hypersensitivity to the study drugs or to drugs with similar chemical structures
* History of severe or multiple allergies
* Treatment with any other investigational drug within 3 months before trial entry
* Progressive fatal disease
* History of drug or alcohol abuse in the past 2 years
* Condition after kidney transplantation
* Serum potassium > 5.5 mmol/L
* Pregnancy or breast feeding
* Sexually active woman of childbearing age not practicing a highly effective method of birth control as defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, sexual abstinence or vasectomised partner.
* Acute myocardial infarction, open heart surgery or cerebral event (stroke/TIA) within the previous 3 months
* Any elective surgery during study participation
* Uncontrolled unstable angina pectoris
* Intake of Coumarin or coumarin derived compounds such as phenprocoumon (Marcumar) or warfarin (Coumadin, Warfant)
* Intake of rifampicin or carbamazepine
* HbA1c ≥ 6,5%
* A Body Mass Index of > 35 kg/m²
* CHF NYHA stage III - IV

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Albumin/Creatinine Ratio (UACR) in 24h urine change between Baseline and Visit 4 | up to 14 weeks of study drug intake

SECONDARY OUTCOMES:
24 hour urinary sodium excretion change between Baseline and Visit 4 | after 14 weeks of study drug intake
Fasting cystatin C change between Baseline and V4 | up to 14 weeks of study drug intake
Fasting cGMP change between Baseline and Visit 4 | after 14 weeks of study drug intake
Fasting serum ADMA change between Baseline and V4 | up to 14 weeks of study drug intake
Fasting hsCRP change between Baseline and Visit 4 | up to 14 weeks of study drug intake
Fasting TGF-ß1 change between Baseline and Visit 4 | after 14 weeks of study drug intake
Retinal endothelial function change between Baseline and Visit 4 | up to 14 weeks of study drug intake
Retinal microvascular blood flow change between Baseline and Visit 4 | up to 14 weeks of study drug intake
24h blood pressure measurements change between Baseline and Visit 4 | up to 14 weeks of study drug intake
HbA1c change between Baseline and Visit 4 | up to 14 weeks of study drug intake
Body weight change during study participation | up to 14 weeks of study drug intake
Adverse events during study participation | up to 14 weeks of study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, MD, PhD, Principal Investigator — Profil GmbH Mainz
Locations (1):
- Profil Mainz GmbH & Co. KG, Mainz, Rhineland-Palatinate, Germany